CLINICAL TRIAL: NCT00025129
Title: A Phase I Trial of VNP4010M, A Novel Alkylating Agent for Patients With Advanced or Metastatic Cancer
Brief Title: VNP40101M in Treating Patients With Advanced Solid Tumors or Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vion Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: VION-CLI-011; CDR0000068919 (Registry Identifier: PDQ (Physician Data Query)); NCI-V01-1669
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2004-03

CONDITIONS: Lymphoma; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; small intestine lymphoma; unspecified adult solid tumor, protocol specific; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; primary central nervous system non-Hodgkin lymphoma; intraocular lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Intraocular Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — laromustine

INTERVENTIONS:
Drug: laromustine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of VNP40101M in treating patients who have advanced solid tumors or lymphomas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of VNP40101M in patients with advanced solid tumors or lymphomas.
* Determine the toxic effects of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.
* Determine the anti-tumor effects of this drug in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive VNP40101M IV over 15 minutes on day 1. Treatment repeats every 4 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 1-6 patients receive escalating doses of VNP40101M until the maximum tolerated dose (MTD) is determined. The MTD is defined as the highest dose at which no more than 1 of 6 patients experiences dose-limiting toxicity.

PROJECTED ACCRUAL: Approximately 20-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced and/or metastatic solid tumor or lymphoma for which no curative or standard effective therapy exists
* Measurable or evaluable metastatic disease
* No other hematologic malignancy
* No large pleural, pericardial, or peritoneal effusions
* No requirement for immediate palliative treatment, including surgery
* No symptomatic brain metastases or metastases with substantial edema

  * Asymptomatic brain metastases or primary CNS disease allowed if neurologic deficits are stable

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* At least 3 months

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hematocrit at least 30% (transfusion allowed)
* No active uncontrolled bleeding

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT and AST no greater than 1.5 times ULN (3 times ULN if liver metastases present)
* Alkaline phosphatase no greater than 1.5 times ULN (3 times ULN if liver or bone metastases present)
* PT and aPTT no greater than 1.5 times ULN
* Albumin at least 2.5 g/dL

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* Ejection fraction at least 45%
* No active heart disease
* No myocardial infarction within the past 3 months
* No symptomatic coronary artery disease
* No arrhythmias requiring medication
* No uncontrolled congestive heart failure

Pulmonary:

* DLCO and FEV_1 at least 60% of predicted
* No dyspnea with minimal to moderate exertion

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* HIV negative
* No active infection
* Persistent stable chronic toxic effects from prior therapy allowed if no greater than grade 1
* No bleeding diathesis (e.g., active peptic ulcer disease)

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior biologic agents and recovered
* At least 6 months since prior high-dose chemotherapy regimen with stem cell support

Chemotherapy:

* See Biologic therapy
* At least 3 weeks since prior cytotoxic agents (6 weeks for nitrosoureas or mitomycin) and recovered

Endocrine therapy:

* At least 2 weeks since prior hormonal therapy and recovered

Radiotherapy:

* At least 3 weeks since prior radiotherapy and recovered

Surgery:

* See Disease Characteristics
* At least 2 weeks since prior surgery and recovered

Other:

* No other concurrent standard therapy for cancer
* No other concurrent investigational agents
* No concurrent disulfiram (Antabuse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-03; Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Sznol, MD, Study Chair — Vion Pharmaceuticals
Locations (3):
- United States (3):
  - Arizona Clinical Research Center, Tucson, Arizona
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Veterans Affairs Medical Center - West Haven, West Haven, Connecticut